CLINICAL TRIAL: NCT06085105
Title: Caring for Providers to Improve Patient Experience (CPIPE) Study: A Cluster Randomized-controlled Trial to Assess the Impact of the CPIPE Intervention on Person-centered Maternity Care
Brief Title: Caring for Providers to Improve Patient Experience (CPIPE) Trial
Acronym: CPIPE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kenya Medical Research Institute (Other); Navrongo Health Research Centre, Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-38843; R01HD110370 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Stress, Psychological; Maternal Health; Healthcare Provider; Adverse Outcomes; Stress, Emotional; Mental Health Issue; Burnout; Burnout, Psychological; Discrimination, Social
Keywords: quality of care; Kenya; providers; mental health; burnout; stress; person-centered care; discrimination; prejudice; unconscious bias
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological; Social Discrimination; Psychological Well-Being; Prejudice; Bias, Implicit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPIPE Intervention arm (Experimental): 1. Training: A two-day training that addresses the following topics: Stress & positive coping mechanisms; Bias awareness and mitigation; Person-centered maternity care; Dealing with difficult situations; and Teamwork and communication. 2. Peer support: Groups for healthcare providers to meet with other healthcare providers of their cadre, to debrief, discuss issues they are facing, brainstorm solutions, and provide support to one another. 3. Leadership engagement: Engagement of County leadership at the onset of the project through a community advisory board to guide and help address sources of stress. 4. Mentorship: mentor-mentee relationships that provide the opportunity to coach less experienced healthcare providers on professional development, work-life balance, clinical skills, career advancement and other topics. 5. Embedded champions: facility champions to lead in organizing and facilitating peer support groups and refreshers at their facilities and serve as role models.
  Interventions: Behavioral: CPIPE Training; Behavioral: Peer support groups; Behavioral: Mentorship; Behavioral: Leadership engagement; Behavioral: Embedded champions
- CPIPE control arm (No Intervention): The control group will not receive the CPIPE intervention during the 12-month data collection period but will maintain their usual facility level activities.

INTERVENTIONS:
Behavioral: CPIPE Training — A two day training covering the following topics: understanding stress & burnout and developing positive coping mechanisms, bias awareness & mitigation, person-centered maternity care mindfulness, dealing with difficult situations, emergency obstetric and neonatal care, teamwork and communication, mentorship and peer support.
  Arms: CPIPE Intervention arm
Behavioral: Peer support groups — Groups for healthcare providers to meet with other healthcare providers of their cadre, and discuss issues they are facing, brainstorm solutions, and provide support to one another.
  Arms: CPIPE Intervention arm
Behavioral: Mentorship — Mentor-mentee relationships that provide the opportunity to coach junior healthcare providers on professional development, work-life balance, clinical skills, career advancement and other topics. Mentors develop their mentorship and leadership skills.
  Arms: CPIPE Intervention arm
Behavioral: Leadership engagement — Engagement of County leadership at the onset of the project through a community advisory board, regular updates of the study and findings, and discussing systemic gaps that impact provider stress and bias.
  Arms: CPIPE Intervention arm
Behavioral: Embedded champions — To facilitate ongoing engagement and sustainability at the facility level, we identified facility champions who lead in organizing and facilitating peer support groups and refreshers at their facilities and serve as role models.
  Arms: CPIPE Intervention arm

SUMMARY:
The activities described in this proposal are aimed at addressing health care provider stress and unconscious bias to improve quality of maternal health care, particularly related to the person-centered dimensions of care-i.e. care that is respectful and responsive to women's needs, preferences, and values. The investigators focus on health provider stress and unconscious bias because they are key drivers of poor-quality care that are often not addressed in interventions designed to improve quality of maternal health care. The investigators plan to (1) test the effectiveness of an intervention that targets provider stress and bias to improve PCMC; (2) assess the cost-effectiveness of CPIPE; (3) examine the mechanisms of impact of CPIPE on PCMC; and (3) assess impact of the CPIPE intervention on distal outcomes including maternal health seeking behavior and maternal and neonatal health.

DETAILED DESCRIPTION:
Poor person-centered maternal care (PCMC) contributes to high maternal mortality and morbidity, directly and indirectly, through lack of, delayed, inadequate, unnecessary, or harmful care. The proposed R01 will test the effectiveness of an intervention that targets provider stress and bias to improve PCMC. The investigators will accomplish this through 3 aims. Aim 1: to assess the effectiveness of the CPIPE intervention on PCMC in Kenya and Ghana. The investigators hypothesize that CPIPE will improve PCMC for all women, and especially for low SES women. The primary outcome is PCMC measured with the PCMC scale through multiple cross-sectional surveys of mothers who gave birth in the preceding 12 weeks in study facilities at baseline (prior to intervention), midline (6 months post-baseline), and endline (12 months post-baseline) (N=2000 at each time point). A sub-aim 1 will assess the cost-effectiveness of CPIPE. Aim 2: to examine the mechanisms of impact of CPIPE on PCMC. The investigators will assess the effect of CPIPE on intermediate outcomes such as provider knowledge, self-efficacy, stress, burnout, and bias levels; and conduct mediation analysis to assess if changes in these outcomes account for the effect of CPIPE on PCMC. Aim 3: to assess impact of the CPIPE intervention on distal outcomes including maternal health seeking behavior and maternal and neonatal health; and examine if changes in PCMC account for these effects.

ELIGIBILITY:
Women's survey

Eligibility criteria

1. Women receiving care at the study facilities.
2. Have given birth within the 12 weeks preceding the data collection.
3. Capable and willing to provide informed consent.
4. Age 15 or above, with individuals aged 15-17 meeting the criteria for emancipated minors as defined by Kenyan or Ghana law (pregnant or parenting, living apart from their parents or guardian; living separately with or without their parents or guardian's consent, regardless of duration; and, controlling their financial affairs regardless of the source of income).

Exclusion criteria

1. Women who are too ill to participate or do not live within a feasible location if interviews are scheduled to be conducted in the community.
2. Women who are younger than 15 years of age.

Provider's cohort

Eligibility criteria

1. Healthcare providers working in maternal health units for at least 6 months at the time of data collection.
2. Capable and willing to provide informed consent.
3. Able and committed to attending the intervention training and follow up activities.
4. Age 18 or above.

Exclusion criteria

1. Healthcare providers planning to no longer be working at the facilities in the next six months, at the time of enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in person-centered maternity care (PCMC) score from baseline to 6 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 6 months
  The PCMC scale is a 30-item scale with 3 sub-scales for dignity and respect, communication and autonomy, and supportive care. Items for each scale are summed to create a score, which is standardized to range from 0 to 100, where higher scores indicate more person-centered care.
Change in person-centered maternity care (PCMC) score from 6 months sustained at 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | 6 months and 12 months
  The PCMC scale is a 30-item scale with 3 sub-scales for dignity and respect, communication and autonomy, and supportive care. Items for each scale are summed to create a score, which is standardized to range from 0 to 100, where higher scores indicate more person-centered care.
Change in person-centered maternity care (PCMC) score from baseline to 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 12 months
  The PCMC scale is a 30-item scale with 3 sub-scales for dignity and respect, communication and autonomy, and supportive care. Items for each scale are summed to create a score, which is standardized to range from 0 to 100, where higher scores indicate more person-centered care.

SECONDARY OUTCOMES:
Change in stress and stress management knowledge and attitude scores from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The stress knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding stress and stress management.
Change in stress and stress management knowledge and attitude scores from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The stress knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding stress and stress management.
Change in stress and stress management knowledge and attitude scores from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The stress knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding stress and stress management.
Change in unconscious bias knowledge and attitude scores from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The unconscious bias knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding unconscious bias.
Change in unconscious bias knowledge and attitude scores from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The unconscious bias knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding unconscious bias.
Change in unconscious bias knowledge and attitude scores from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The unconscious bias knowledge and attitudes score is measured by 10 survey questions with scores ranging from 0 to 10. Higher scores indicate higher knowledge and positive attitudes regarding unconscious bias.
Change in Perceived Stress Scale (PSS) score from baseline to 6 Months, among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  Perceived Stress is measured by the 10-item Cohen Perceived Stress Scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Change in Perceived Stress Scale (PSS) score from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  Perceived Stress is measured by the 10-item Cohen Perceived Stress Scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Change in Perceived Stress Scale (PSS) score from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  Perceived Stress is measured by the 10-item Cohen Perceived Stress Scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Change in Shirom-Melamed Burnout Measure (SMBM) score from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The Shirom-Melamed Burnout Measure is a 14-item scale. Scores range from 1 to 7 with higher scores indicating higher burnout.
Change in Shirom-Melamed Burnout Measure (SMBM) score from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The Shirom-Melamed Burnout Measure is a 14-item scale. Scores range from 1 to 7 with higher scores indicating higher burnout.
Change in Shirom-Melamed Burnout Measure (SMBM) score from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The Shirom-Melamed Burnout Measure is a 14-item scale. Scores range from 1 to 7 with higher scores indicating higher burnout.
Change in bias awareness and mitigation scores from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The scale is composed of the following 3 subscales: a 9-item Bias Awareness subscale; and a 7-item Bias Mitigation Self-Efficacy sub-scale; and 7-item Bias mitigation subscale.
Change in bias awareness and mitigation scores from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The scale is composed of the following 3 subscales: a 9-item Bias Awareness subscale; and a 7-item Bias Mitigation Self-Efficacy sub-scale; and 7-item Bias mitigation subscale.
Change in bias awareness and mitigation scores from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The scale is composed of the following 3 subscales: a 9-item Bias Awareness subscale; and a 7-item Bias Mitigation Self-Efficacy sub-scale; and 7-item Bias mitigation subscale.
Change in explicit bias scores from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The explicit bias scores are from responses to a vignette and range from 4 to 28. Higher scores indicate more explicit bias.
Change in explicit bias scores from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The explicit bias scores are from responses to a vignette and range from 4 to 28. Higher scores indicate more explicit bias.
Change in explicit bias scores from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The explicit bias scores are from responses to a vignette and range from 4 to 28. Higher scores indicate more explicit bias.
Change in supportive environment score from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  Survey questions to assess support from leadership, superiors and colleagues, indicating a more supportive and enabling environment.
Change in supportive environment score from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  Survey questions to assess support from leadership, superiors and colleagues, indicating a more supportive and enabling environment.
Change in supportive environment score from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  Survey questions to assess support from leadership, superiors and colleagues, indicating a more supportive and enabling environment.
Change in self-reported PCMC provision scores from baseline to 6 months among providers in intervention facilities compared to those in control facilities. | Baseline and 6 months
  The 9-item provider reported PCMC scale ranges from 0 to 27 with higher scores indicating higher PCMC provision.
Change in self-reported PCMC provision scores from 6 months sustained at 12 months among providers in intervention facilities compared to those in control facilities. | 6 months and 12 months
  The 9-item provider reported PCMC scale ranges from 0 to 27 with higher scores indicating higher PCMC provision.
Change in self-reported PCMC provision scores from baseline to 12 months among providers in intervention facilities compared to those in control facilities. | Baseline and 12 months
  The 9-item provider reported PCMC scale ranges from 0 to 27 with higher scores indicating higher PCMC provision.
Change in postnatal care utilization from baseline to 6 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 6 months
  Survey questions on receipt and timing of postnatal care
Change in postnatal care utilization from 6 months sustained at 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | 6 months and 12 months
  Survey questions on receipt and timing of postnatal care
Change in postnatal care utilization from baseline to 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 12 months
  Survey questions on receipt and timing of postnatal care
Change in breastfeeding rates from baseline to 6 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 6 months
  Survey questions on breastfeeding initiation, exclusive breastfeeding, and duration of breastfeeding
Change in breastfeeding rates from 6 months sustained at 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | 6 months and 12 months
  Survey questions on breastfeeding initiation, exclusive breastfeeding, and duration of breastfeeding
Change in breastfeeding rates from baseline to 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 12 months
  Survey questions on breastfeeding initiation, exclusive breastfeeding, and duration of breastfeeding
Change in post-partum depression rates from baseline to 6 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 6 months
  10-item Edinburgh Perinatal/Postnatal Depression Scale (EPDS). Scores range from 0 to 30 with higher scores indicating more severe depression
Change in post-partum depression rates from 6 months sustained at 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | 6 months and 12 months
  10-item Edinburgh Perinatal/Postnatal Depression Scale (EPDS). Scores range from 0 to 30 with higher scores indicating more severe depression
Change in post-partum depression rates from baseline to 12 months among women who give birth in intervention facilities compared to those who give birth in control facilities. | Baseline and 12 months
  10-item Edinburgh Perinatal/Postnatal Depression Scale (EPDS). Scores range from 0 to 30 with higher scores indicating more severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Patience Afulani, PhD, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Upper East and North East regions health facilities, Navrongo, Ghana
- Migori and Homabay Counties health facilities, Migori, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afulani PA, Diamond-Smith N, Golub G, Sudhinaraset M. Development of a tool to measure person-centered maternity care in developing settings: validation in a rural and urban Kenyan population. Reprod Health. 2017 Sep 22;14(1):118. doi: 10.1186/s12978-017-0381-7. PMID 28938885
- [Background] Alkema L, Chou D, Hogan D, Zhang S, Moller AB, Gemmill A, Fat DM, Boerma T, Temmerman M, Mathers C, Say L; United Nations Maternal Mortality Estimation Inter-Agency Group collaborators and technical advisory group. Global, regional, and national levels and trends in maternal mortality between 1990 and 2015, with scenario-based projections to 2030: a systematic analysis by the UN Maternal Mortality Estimation Inter-Agency Group. Lancet. 2016 Jan 30;387(10017):462-74. doi: 10.1016/S0140-6736(15)00838-7. Epub 2015 Nov 13. PMID 26584737
- [Background] Friberg IK, Kinney MV, Lawn JE, Kerber KJ, Odubanjo MO, Bergh AM, Walker N, Weissman E, Chopra M, Black RE; Science in Action: Saving the lives of Africa's Mothers, Newborns, and Children working group; Axelson H, Cohen B, Coovadia H, Diab R, Nkrumah F. Sub-Saharan Africa's mothers, newborns, and children: how many lives could be saved with targeted health interventions? PLoS Med. 2010 Jun 21;7(6):e1000295. doi: 10.1371/journal.pmed.1000295. PMID 20574515
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Gabrysch S, Campbell OM. Still too far to walk: literature review of the determinants of delivery service use. BMC Pregnancy Childbirth. 2009 Aug 11;9:34. doi: 10.1186/1471-2393-9-34. PMID 19671156
- [Background] Moyer CA, Mustafa A. Drivers and deterrents of facility delivery in sub-Saharan Africa: a systematic review. Reprod Health. 2013 Aug 20;10:40. doi: 10.1186/1742-4755-10-40. PMID 23962135
- [Background] van den Broek NR, Graham WJ. Quality of care for maternal and newborn health: the neglected agenda. BJOG. 2009 Oct;116(Suppl 1):18-21. doi: 10.1111/j.1471-0528.2009.02333.x. PMID 19740165
- [Background] Graham WJ, McCaw-Binns A, Munjanja S. Translating coverage gains into health gains for all women and children: the quality care opportunity. PLoS Med. 2013;10(1):e1001368. doi: 10.1371/journal.pmed.1001368. Epub 2013 Jan 15. PMID 23335862
- [Background] Koblinsky M, Moyer CA, Calvert C, Campbell J, Campbell OM, Feigl AB, Graham WJ, Hatt L, Hodgins S, Matthews Z, McDougall L, Moran AC, Nandakumar AK, Langer A. Quality maternity care for every woman, everywhere: a call to action. Lancet. 2016 Nov 5;388(10057):2307-2320. doi: 10.1016/S0140-6736(16)31333-2. Epub 2016 Sep 16. PMID 27642018
- [Background] Anwar I, Kalim N, Koblinsky M. Quality of obstetric care in public-sector facilities and constraints to implementing emergency obstetric care services: evidence from high- and low-performing districts of Bangladesh. J Health Popul Nutr. 2009 Apr;27(2):139-55. doi: 10.3329/jhpn.v27i2.3327. PMID 19489412
- [Background] Donabedian A. The quality of care. How can it be assessed? JAMA. 1988 Sep 23-30;260(12):1743-8. doi: 10.1001/jama.260.12.1743. PMID 3045356
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Bohren MA, Hunter EC, Munthe-Kaas HM, Souza JP, Vogel JP, Gulmezoglu AM. Facilitators and barriers to facility-based delivery in low- and middle-income countries: a qualitative evidence synthesis. Reprod Health. 2014 Sep 19;11(1):71. doi: 10.1186/1742-4755-11-71. PMID 25238684
- [Background] Bohren MA, Vogel JP, Hunter EC, Lutsiv O, Makh SK, Souza JP, Aguiar C, Saraiva Coneglian F, Diniz AL, Tuncalp O, Javadi D, Oladapo OT, Khosla R, Hindin MJ, Gulmezoglu AM. The Mistreatment of Women during Childbirth in Health Facilities Globally: A Mixed-Methods Systematic Review. PLoS Med. 2015 Jun 30;12(6):e1001847; discussion e1001847. doi: 10.1371/journal.pmed.1001847. eCollection 2015 Jun. PMID 26126110
- [Background] Afulani PA, Kirumbi L, Lyndon A. What makes or mars the facility-based childbirth experience: thematic analysis of women's childbirth experiences in western Kenya. Reprod Health. 2017 Dec 29;14(1):180. doi: 10.1186/s12978-017-0446-7. PMID 29284490
- [Background] Odiase O, Akinyi B, Kinyua J, Afulani P. Community Perceptions of Person-Centered Maternity Care in Migori County, Kenya. Front Glob Womens Health. 2021 Oct 8;2:668405. doi: 10.3389/fgwh.2021.668405. eCollection 2021. PMID 34816219
- [Background] Afulani PA, Phillips B, Aborigo RA, Moyer CA. Person-centred maternity care in low-income and middle-income countries: analysis of data from Kenya, Ghana, and India. Lancet Glob Health. 2019 Jan;7(1):e96-e109. doi: 10.1016/S2214-109X(18)30403-0. PMID 30554766
- [Background] Afulani PA, Sayi TS, Montagu D. Predictors of person-centered maternity care: the role of socioeconomic status, empowerment, and facility type. BMC Health Serv Res. 2018 May 11;18(1):360. doi: 10.1186/s12913-018-3183-x. PMID 29751805
- [Background] Andersen HM. "Villagers": differential treatment in a Ghanaian hospital. Soc Sci Med. 2004 Nov;59(10):2003-12. doi: 10.1016/j.socscimed.2004.03.005. PMID 15351468
- [Background] Atinga RA, Bawole JN, Nang-Beifubah A. 'Some patients are more equal than others': Patient-centred care differential in two-tier inpatient ward hospitals in Ghana. Patient Educ Couns. 2016 Mar;99(3):370-377. doi: 10.1016/j.pec.2015.09.008. Epub 2015 Oct 9. PMID 26475729
- [Background] Bohren MA, Mehrtash H, Fawole B, Maung TM, Balde MD, Maya E, Thwin SS, Aderoba AK, Vogel JP, Irinyenikan TA, Adeyanju AO, Mon NO, Adu-Bonsaffoh K, Landoulsi S, Guure C, Adanu R, Diallo BA, Gulmezoglu AM, Soumah AM, Sall AO, Tuncalp O. How women are treated during facility-based childbirth in four countries: a cross-sectional study with labour observations and community-based surveys. Lancet. 2019 Nov 9;394(10210):1750-1763. doi: 10.1016/S0140-6736(19)31992-0. Epub 2019 Oct 8. PMID 31604660
- [Background] Miller S, Abalos E, Chamillard M, Ciapponi A, Colaci D, Comande D, Diaz V, Geller S, Hanson C, Langer A, Manuelli V, Millar K, Morhason-Bello I, Castro CP, Pileggi VN, Robinson N, Skaer M, Souza JP, Vogel JP, Althabe F. Beyond too little, too late and too much, too soon: a pathway towards evidence-based, respectful maternity care worldwide. Lancet. 2016 Oct 29;388(10056):2176-2192. doi: 10.1016/S0140-6736(16)31472-6. Epub 2016 Sep 16. PMID 27642019
- [Background] Fahy K. What is woman-centred care and why does it matter? Women Birth. 2012 Dec;25(4):149-51. doi: 10.1016/j.wombi.2012.10.005. No abstract available. PMID 23177665
- [Background] Bohren MA, Hofmeyr GJ, Sakala C, Fukuzawa RK, Cuthbert A. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2017 Jul 6;7(7):CD003766. doi: 10.1002/14651858.CD003766.pub6. PMID 28681500
- [Background] Doyle C, Lennox L, Bell D. A systematic review of evidence on the links between patient experience and clinical safety and effectiveness. BMJ Open. 2013 Jan 3;3(1):e001570. doi: 10.1136/bmjopen-2012-001570. PMID 23293244
- [Background] Oliveira VC, Refshauge KM, Ferreira ML, Pinto RZ, Beckenkamp PR, Negrao Filho RF, Ferreira PH. Communication that values patient autonomy is associated with satisfaction with care: a systematic review. J Physiother. 2012;58(4):215-29. doi: 10.1016/S1836-9553(12)70123-6. PMID 23177224
- [Background] Afulani PA, Aborigo RA, Walker D, Moyer CA, Cohen S, Williams J. Can an integrated obstetric emergency simulation training improve respectful maternity care? Results from a pilot study in Ghana. Birth. 2019 Sep;46(3):523-532. doi: 10.1111/birt.12418. Epub 2019 Jan 24. PMID 30680785
- [Background] Afulani PA, Buback L, Essandoh F, Kinyua J, Kirumbi L, Cohen CR. Quality of antenatal care and associated factors in a rural county in Kenya: an assessment of service provision and experience dimensions. BMC Health Serv Res. 2019 Oct 7;19(1):684. doi: 10.1186/s12913-019-4476-4. PMID 31590662
- [Background] Montagu D, Landrian A, Kumar V, Phillips BS, Singhal S, Mishra S, Singh S, Cotter SY, Singh VP, Kajal F, Sudhinaraset M. Patient-experience during delivery in public health facilities in Uttar Pradesh, India. Health Policy Plan. 2019 Oct 1;34(8):574-581. doi: 10.1093/heapol/czz067. PMID 31419287
- [Background] Bohren MA, Vogel JP, Tuncalp O, Fawole B, Titiloye MA, Olutayo AO, Oyeniran AA, Ogunlade M, Metiboba L, Osunsan OR, Idris HA, Alu FE, Oladapo OT, Gulmezoglu AM, Hindin MJ. "By slapping their laps, the patient will know that you truly care for her": A qualitative study on social norms and acceptability of the mistreatment of women during childbirth in Abuja, Nigeria. SSM Popul Health. 2016 Dec;2:640-655. doi: 10.1016/j.ssmph.2016.07.003. PMID 28345016
- [Background] Burrowes S, Holcombe SJ, Jara D, Carter D, Smith K. Midwives' and patients' perspectives on disrespect and abuse during labor and delivery care in Ethiopia: a qualitative study. BMC Pregnancy Childbirth. 2017 Aug 22;17(1):263. doi: 10.1186/s12884-017-1442-1. PMID 28830383
- [Background] Warren CE, Njue R, Ndwiga C, Abuya T. Manifestations and drivers of mistreatment of women during childbirth in Kenya: implications for measurement and developing interventions. BMC Pregnancy Childbirth. 2017 Mar 28;17(1):102. doi: 10.1186/s12884-017-1288-6. PMID 28351350
- [Background] Rominski SD, Lori J, Nakua E, Dzomeku V, Moyer CA. When the baby remains there for a long time, it is going to die so you have to hit her small for the baby to come out": justification of disrespectful and abusive care during childbirth among midwifery students in Ghana. Health Policy Plan. 2017 Mar 1;32(2):215-224. doi: 10.1093/heapol/czw114. PMID 28207054
- [Background] Jewkes R, Abrahams N, Mvo Z. Why do nurses abuse patients? Reflections from South African obstetric services. Soc Sci Med. 1998 Dec;47(11):1781-95. doi: 10.1016/s0277-9536(98)00240-8. PMID 9877348
- [Background] Sen G, Reddy B, Iyer A. Beyond measurement: the drivers of disrespect and abuse in obstetric care. Reprod Health Matters. 2018;26(53):6-18. doi: 10.1080/09688080.2018.1508173. Epub 2018 Sep 7. PMID 30189791
- [Background] Afulani PA, Buback L, Kelly AM, Kirumbi L, Cohen CR, Lyndon A. Providers' perceptions of communication and women's autonomy during childbirth: a mixed methods study in Kenya. Reprod Health. 2020 Jun 3;17(1):85. doi: 10.1186/s12978-020-0909-0. PMID 32493424
- [Background] Buback L, Kinyua J, Akinyi B, Walker D, Afulani PA. Provider perceptions of lack of supportive care during childbirth: A mixed methods study in Kenya. Health Care Women Int. 2022 Sep;43(9):1062-1083. doi: 10.1080/07399332.2021.1961776. Epub 2021 Sep 17. PMID 34534038
- [Background] Jewkes R, Penn-Kekana L. Mistreatment of Women in Childbirth: Time for Action on This Important Dimension of Violence against Women. PLoS Med. 2015 Jun 30;12(6):e1001849. doi: 10.1371/journal.pmed.1001849. eCollection 2015 Jun. No abstract available. PMID 26126175
- [Background] Freedman LP, Kruk ME. Disrespect and abuse of women in childbirth: challenging the global quality and accountability agendas. Lancet. 2014 Sep 20;384(9948):e42-4. doi: 10.1016/S0140-6736(14)60859-X. Epub 2014 Jun 22. No abstract available. PMID 24965825
- [Background] Downe S, Lawrie TA, Finlayson K, Oladapo OT. Effectiveness of respectful care policies for women using routine intrapartum services: a systematic review. Reprod Health. 2018 Feb 6;15(1):23. doi: 10.1186/s12978-018-0466-y. PMID 29409519
- [Background] Ratcliffe HL, Sando D, Lyatuu GW, Emil F, Mwanyika-Sando M, Chalamilla G, Langer A, McDonald KP. Mitigating disrespect and abuse during childbirth in Tanzania: an exploratory study of the effects of two facility-based interventions in a large public hospital. Reprod Health. 2016 Jul 18;13(1):79. doi: 10.1186/s12978-016-0187-z. PMID 27424608
- [Background] Abuya T, Ndwiga C, Ritter J, Kanya L, Bellows B, Binkin N, Warren CE. The effect of a multi-component intervention on disrespect and abuse during childbirth in Kenya. BMC Pregnancy Childbirth. 2015 Sep 22;15:224. doi: 10.1186/s12884-015-0645-6. PMID 26394616
- [Background] Afulani PA, Kelly AM, Buback L, Asunka J, Kirumbi L, Lyndon A. Providers' perceptions of disrespect and abuse during childbirth: a mixed-methods study in Kenya. Health Policy Plan. 2020 Jun 1;35(5):577-586. doi: 10.1093/heapol/czaa009. PMID 32154878
- [Background] Afulani PA, Aborigo RA, Nutor JJ, Okiring J, Kuwolamo I, Ogolla BA, Oboke EN, Dorzie JBK, Odiase OJ, Steinauer J, Walker D. Self-reported provision of person-centred maternity care among providers in Kenya and Ghana: scale validation and examination of associated factors. BMJ Glob Health. 2021 Nov;6(12):e007415. doi: 10.1136/bmjgh-2021-007415. PMID 34853033
- [Background] Afulani PA, Ongeri L, Kinyua J, Temmerman M, Mendes WB, Weiss SJ. Psychological and physiological stress and burnout among maternity providers in a rural county in Kenya: individual and situational predictors. BMC Public Health. 2021 Mar 6;21(1):453. doi: 10.1186/s12889-021-10453-0. PMID 33676479
- [Background] WHO. PMNCH Fact Sheet: Maternal mortality. Published 2011. Accessed July 16, 2013. http://www.who.int/pmnch/media/press_materials/fs/fs_mdg5_maternalmortality/en/index.html
- [Background] WHO. Making pregnancy safer: the critical role of the skilled attendant. Jt Statement WHO ICM FIGO Geneva. Published online 2004.
- [Background] WHO. Global Health Observatory Data Repository, MDG 5: Maternal health: Published 2013. Accessed September 5, 2013. http://apps.who.int/gho/data/node.main.REPWOMEN39
- [Background] March of Dimes, PMNCH, Save the Children. Born Too Soon: The Global Action Report on Preterm Birth. Eds CP Howson, MV Kinney, JE Lawn. Published online 2012.
- [Background] UNICEF. Antenatal care: Joint UNICEF/WHO database 2021 of skilled health personnel, based on population based national household survey data and routine health systems. UNICEF DATA. Published 2021. Accessed November 3, 2021. https://data.unicef.org/topic/maternal-health/antenatal-care/
- [Background] UNICEF. Delivery care: Joint UNICEF/WHO database 2021 of skilled health personnel, based on population based national household survey data and routine health systems. UNICEF DATA. Published 2021. Accessed November 1, 2021. https://data.unicef.org/topic/maternal-health/delivery-care/
- [Background] GSS GSS, GHS GHS, ICF. Ghana Maternal Health Survey 2017. Published online August 1, 2018. Accessed December 29, 2019. https://www.dhsprogram.com/publications/publication-FR340-Other-Final-Reports.cfm
- [Background] Kenya National Bureau of Statistics, Ministry of Health, National AIDS Control Council, Kenya Medical Research Institute, National Council for Population and Development, Nairobi, Kenya, and The DHS Program, ICF International, Rockville, Maryland, USA. The DHS Program - Kenya: DHS, 2014 - Final Report (English).; 2015. Accessed February 18, 2016. http://dhsprogram.com/publications/publication-FR308-DHS-Final-Reports.cfm
- [Background] Leavitt M. Medscape's response to the Institute of Medicine Report: Crossing the quality chasm: a new health system for the 21st century. MedGenMed. 2001 Mar 5;3(2):2. No abstract available. PMID 11549951
- [Background] WHO. Prevention and elimination of disrespect and abuse during childbirth. WHO. Published 2014. Accessed April 4, 2017. http://www.who.int/reproductivehealth/topics/maternal_perinatal/statement-childbirth/en/
- [Background] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] White Ribbon Alliance. Respectful Maternity Care: The Universal Rights of Childbearing Women (Full charter). Published 2011. Accessed March 28, 2017. http://www.healthpolicyproject.com/index.cfm?ID=publications&get=pubID&pubID=46
- [Background] Filby A, McConville F, Portela A. What Prevents Quality Midwifery Care? A Systematic Mapping of Barriers in Low and Middle Income Countries from the Provider Perspective. PLoS One. 2016 May 2;11(5):e0153391. doi: 10.1371/journal.pone.0153391. eCollection 2016. PMID 27135248
- [Background] Fauveau V, Sherratt DR, de Bernis L. Human resources for maternal health: multi-purpose or specialists? Hum Resour Health. 2008 Sep 30;6:21. doi: 10.1186/1478-4491-6-21. PMID 18826600
- [Background] McEwen BS. Stressed or stressed out: what is the difference? J Psychiatry Neurosci. 2005 Sep;30(5):315-8. PMID 16151535
- [Background] Public Health England. Interventions to prevent burnout in high risk individuals: evidence review - Publications - GOV.UK. Published 2016. Accessed October 26, 2016. https://www.gov.uk/government/publications/interventions-to-prevent-burnout-in-high-risk-individuals-evidence-review
- [Background] Halbesleben JRB, ed. Handbook of Stress and Burnout in Health Care. 3 edition. Nova Science Pub Inc; 2008.
- [Background] Wallace JE, Lemaire JB, Ghali WA. Physician wellness: a missing quality indicator. Lancet. 2009 Nov 14;374(9702):1714-21. doi: 10.1016/S0140-6736(09)61424-0. PMID 19914516
- [Background] Klein J, Grosse Frie K, Blum K, von dem Knesebeck O. Burnout and perceived quality of care among German clinicians in surgery. Int J Qual Health Care. 2010 Dec;22(6):525-30. doi: 10.1093/intqhc/mzq056. Epub 2010 Oct 8. PMID 20935011
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] Shanafelt TD, Sloan JA, Habermann TM. The well-being of physicians. Am J Med. 2003 Apr 15;114(6):513-9. doi: 10.1016/s0002-9343(03)00117-7. No abstract available. PMID 12727590
- [Background] Afulani PA, Gyamerah AO, Nutor JJ, Laar A, Aborigo RA, Malechi H, Sterling M, Awoonor-Williams JK. Inadequate preparedness for response to COVID-19 is associated with stress and burnout among healthcare workers in Ghana. PLoS One. 2021 Apr 16;16(4):e0250294. doi: 10.1371/journal.pone.0250294. eCollection 2021. PMID 33861808
- [Background] Afulani PA, Nutor JJ, Agbadi P, Gyamerah AO, Musana J, Aborigo RA, Odiase O, Getahun M, Ongeri L, Malechi H, Madadi MO, Arhinful B, Kelly AM, Awoonor-Williams JK. Job satisfaction among healthcare workers in Ghana and Kenya during the COVID-19 pandemic: Role of perceived preparedness, stress, and burnout. PLOS Glob Public Health. 2021 Oct 13;1(10):e0000022. doi: 10.1371/journal.pgph.0000022. eCollection 2021. PMID 36962085
- [Background] Pappa S, Ntella V, Giannakas T, Giannakoulis VG, Papoutsi E, Katsaounou P. Prevalence of depression, anxiety, and insomnia among healthcare workers during the COVID-19 pandemic: A systematic review and meta-analysis. Brain Behav Immun. 2020 Aug;88:901-907. doi: 10.1016/j.bbi.2020.05.026. Epub 2020 May 8. PMID 32437915
- [Background] Busch IM, Moretti F, Mazzi M, Wu AW, Rimondini M. What We Have Learned from Two Decades of Epidemics and Pandemics: A Systematic Review and Meta-Analysis of the Psychological Burden of Frontline Healthcare Workers. Psychother Psychosom. 2021;90(3):178-190. doi: 10.1159/000513733. Epub 2021 Feb 1. PMID 33524983
- [Background] Li Y, Scherer N, Felix L, Kuper H. Prevalence of depression, anxiety and post-traumatic stress disorder in health care workers during the COVID-19 pandemic: A systematic review and meta-analysis. PLoS One. 2021 Mar 10;16(3):e0246454. doi: 10.1371/journal.pone.0246454. eCollection 2021. PMID 33690641
- [Background] Blair IV, Steiner JF, Havranek EP. Unconscious (implicit) bias and health disparities: where do we go from here? Perm J. 2011 Spring;15(2):71-8. doi: 10.7812/TPP/11.979. PMID 21841929
- [Background] Mendes WB, Koslov K. Brittle smiles: positive biases toward stigmatized and outgroup targets. J Exp Psychol Gen. 2013 Aug;142(3):923-33. doi: 10.1037/a0029663. Epub 2012 Aug 13. PMID 22889160
- [Background] UNC Executive Development. The Real Effects of Unconscious Bias in the Workplace. Published 2015. Accessed October 26, 2016. http://execdev.kenan-flagler.unc.edu/blog/the-real-effects-of-unconscious-bias-in-the-workplace-0
- [Background] Nosek BA, Ranganath KA, Smith CT, et al. Pervasiveness and Correlates of Implicit Attitudes and Stereotypes. Published online 2007. Accessed December 8, 2016. https://dash.harvard.edu/handle/1/2958438
- [Background] Green AR, Carney DR, Pallin DJ, Ngo LH, Raymond KL, Iezzoni LI, Banaji MR. Implicit bias among physicians and its prediction of thrombolysis decisions for black and white patients. J Gen Intern Med. 2007 Sep;22(9):1231-8. doi: 10.1007/s11606-007-0258-5. Epub 2007 Jun 27. PMID 17594129
- [Background] Cooper LA, Roter DL, Carson KA, Beach MC, Sabin JA, Greenwald AG, Inui TS. The associations of clinicians' implicit attitudes about race with medical visit communication and patient ratings of interpersonal care. Am J Public Health. 2012 May;102(5):979-87. doi: 10.2105/AJPH.2011.300558. Epub 2012 Mar 15. PMID 22420787
- [Background] Sabin JA, Greenwald AG. The influence of implicit bias on treatment recommendations for 4 common pediatric conditions: pain, urinary tract infection, attention deficit hyperactivity disorder, and asthma. Am J Public Health. 2012 May;102(5):988-95. doi: 10.2105/AJPH.2011.300621. Epub 2012 Mar 15. PMID 22420817
- [Background] Sudhinaraset M, Beyeler N, Barge S, Diamond-Smith N. Decision-making for delivery location and quality of care among slum-dwellers: a qualitative study in Uttar Pradesh, India. BMC Pregnancy Childbirth. 2016 Jul 7;16:148. doi: 10.1186/s12884-016-0942-8. PMID 27387024
- [Background] Diamond-Smith N, Treleaven E, Murthy N, Sudhinaraset M. Women's empowerment and experiences of mistreatment during childbirth in facilities in Lucknow, India: results from a cross-sectional study. BMC Pregnancy Childbirth. 2017 Nov 8;17(Suppl 2):335. doi: 10.1186/s12884-017-1501-7. PMID 29143668
- [Background] Leape LL, Shore MF, Dienstag JL, Mayer RJ, Edgman-Levitan S, Meyer GS, Healy GB. Perspective: a culture of respect, part 1: the nature and causes of disrespectful behavior by physicians. Acad Med. 2012 Jul;87(7):845-52. doi: 10.1097/ACM.0b013e318258338d. PMID 22622217
- [Background] Leape LL, Shore MF, Dienstag JL, Mayer RJ, Edgman-Levitan S, Meyer GS, Healy GB. Perspective: a culture of respect, part 2: creating a culture of respect. Acad Med. 2012 Jul;87(7):853-8. doi: 10.1097/ACM.0b013e3182583536. PMID 22622219
- [Background] Afulani PA, Ogolla BA, Oboke EN, Ongeri L, Weiss SJ, Lyndon A, Mendes WB. Understanding disparities in person-centred maternity care: the potential role of provider implicit and explicit bias. Health Policy Plan. 2021 Apr 21;36(3):298-311. doi: 10.1093/heapol/czaa190. PMID 33491086
- [Background] Rubashkin N, Warnock R, Diamond-Smith N. A systematic review of person-centered care interventions to improve quality of facility-based delivery. Reprod Health. 2018 Oct 10;15(1):169. doi: 10.1186/s12978-018-0588-2. PMID 30305129
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Glanz K, Rimer KB. Theory at a Glance: A Guide for Health Promotion Practice. National Cancer Institute, National Institutes of Health, U.S. Department of Health and Human Services. NIH Pub. No. 97-3896. Washington, DC: NIH.; 1997.
- [Background] San Francisco Department of Public Health. Trauma Informed Systems Initiative 2014 Year in Review. Published online 2015. http://www.leapsf.org/pdf/Trauma-Informed-Systems-Initative-2014.pdf
- [Background] Bloom SL. Organizational Stress and Trauma-Informed Services. In: Levin BL, Becker MA, eds. A Public Health Perspective of Women's Mental Health. Springer New York; 2010:295-311. doi:10.1007/978-1-4419-1526-9_15
- [Background] Cohen SR, Cragin L, Rizk M, Hanberg A, Walker DM. PartoPantsTM: The High-Fidelity, Low-Tech Birth Simulator. Clin Simul Nurs. 2011;7(1):e11-e18. doi:10.1016/j.ecns.2009.11.012
- [Background] Devine PG, Forscher PS, Austin AJ, Cox WT. Long-term reduction in implicit race bias: A prejudice habit-breaking intervention. J Exp Soc Psychol. 2012 Nov;48(6):1267-1278. doi: 10.1016/j.jesp.2012.06.003. PMID 23524616
- [Background] Okonofua JA, Saadatian K, Ocampo J, Ruiz M, Oxholm PD. A scalable empathic supervision intervention to mitigate recidivism from probation and parole. Proc Natl Acad Sci U S A. 2021 Apr 6;118(14):e2018036118. doi: 10.1073/pnas.2018036118. PMID 33782121
- [Background] Okonofua JA, Perez AD, Darling-Hammond S. When policy and psychology meet: Mitigating the consequences of bias in schools. Sci Adv. 2020 Oct 16;6(42):eaba9479. doi: 10.1126/sciadv.aba9479. Print 2020 Oct. PMID 33067225
- [Background] Afulani PA, Dyer J, Calkins K, Aborigo RA, Mcnally B, Cohen SR. Provider knowledge and perceptions following an integrated simulation training on emergency obstetric and neonatal care and respectful maternity care: A mixed-methods study in Ghana. Midwifery. 2020 Jun;85:102667. doi: 10.1016/j.midw.2020.102667. Epub 2020 Feb 19. PMID 32114318
- [Background] Moyer CA, McNally B, Aborigo RA, Williams JEO, Afulani P. Providing respectful maternity care in northern Ghana: A mixed-methods study with maternity care providers. Midwifery. 2021 Mar;94:102904. doi: 10.1016/j.midw.2020.102904. Epub 2020 Dec 11. PMID 33341537
- [Background] Health Policy Project. Kenya County Health Fact Sheets. Published online 2015.
- [Background] Ghana Health Service. Regional health Directorate-Upper East Region. 2018 Annual Report.
- [Background] Ghana Health Service. Upper East Regional Profile-2021.
- [Background] North East Regional Health Directorate. Midyear Performance Review Report 2021.
- [Background] Kruk ME, Leslie HH, Verguet S, Mbaruku GM, Adanu RMK, Langer A. Quality of basic maternal care functions in health facilities of five African countries: an analysis of national health system surveys. Lancet Glob Health. 2016 Nov;4(11):e845-e855. doi: 10.1016/S2214-109X(16)30180-2. Epub 2016 Sep 23. PMID 27670090
- [Background] Walker D, Otieno P, Butrick E, Namazzi G, Achola K, Merai R, Otare C, Mubiri P, Ghosh R, Santos N, Miller L, Sloan NL, Waiswa P; Preterm Birth Initiative Kenya and Uganda Implementation Research Collaborative. Effect of a quality improvement package for intrapartum and immediate newborn care on fresh stillbirth and neonatal mortality among preterm and low-birthweight babies in Kenya and Uganda: a cluster-randomised facility-based trial. Lancet Glob Health. 2020 Aug;8(8):e1061-e1070. doi: 10.1016/S2214-109X(20)30232-1. PMID 32710862
- [Background] Rossi PH, Lipsey MW, Freeman HE. Evaluation: A Systematic Approach. 7th Ed. Thousand Oaks, CA: Sage Publications, Inc.; 2004:68-81.
- [Background] Afulani PA, Altman MR, Castillo E, Bernal N, Jones L, Camara TL, Carrasco Z, Williams S, Sudhinaraset M, Kuppermann M. Development of the person-centered prenatal care scale for people of color. Am J Obstet Gynecol. 2021 Oct;225(4):427.e1-427.e13. doi: 10.1016/j.ajog.2021.04.216. Epub 2021 Apr 20. PMID 33862014
- [Background] Carroll C, Patterson M, Wood S, Booth A, Rick J, Balain S. A conceptual framework for implementation fidelity. Implement Sci. 2007 Nov 30;2:40. doi: 10.1186/1748-5908-2-40. PMID 18053122
- [Background] Breitenstein SM, Gross D, Garvey CA, Hill C, Fogg L, Resnick B. Implementation fidelity in community-based interventions. Res Nurs Health. 2010 Apr;33(2):164-73. doi: 10.1002/nur.20373. PMID 20198637
- [Background] Proctor EK, Powell BJ, Baumann AA, Hamilton AM, Santens RL. Writing implementation research grant proposals: ten key ingredients. Implement Sci. 2012 Oct 12;7:96. doi: 10.1186/1748-5908-7-96. PMID 23062065
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gerber M, Colledge F, Mucke M, Schilling R, Brand S, Ludyga S. Psychometric properties of the Shirom-Melamed Burnout Measure (SMBM) among adolescents: results from three cross-sectional studies. BMC Psychiatry. 2018 Aug 25;18(1):266. doi: 10.1186/s12888-018-1841-5. PMID 30144799
- [Background] Bower KM, Kramer B, Warren N, Ahmed S, Callaghan-Koru J, Stierman E, Wilson C, Lawson S, Creanga AA. Development of an instrument to measure awareness and mitigation of bias in maternal healthcare. Am J Obstet Gynecol MFM. 2023 Apr;5(4):100872. doi: 10.1016/j.ajogmf.2023.100872. Epub 2023 Jan 20. PMID 36682457
- [Background] Sudhinaraset M, Landrian A, Afulani PA, Diamond-Smith N, Golub G. Association between person-centered maternity care and newborn complications in Kenya. Int J Gynaecol Obstet. 2020 Jan;148(1):27-34. doi: 10.1002/ijgo.12978. Epub 2019 Oct 9. PMID 31544243
- [Background] Sudhinaraset M, Landrian A, Golub GM, Cotter SY, Afulani PA. Person-centered maternity care and postnatal health: associations with maternal and newborn health outcomes. AJOG Glob Rep. 2021 Feb;1(1):100005. doi: 10.1016/j.xagr.2021.100005. PMID 33889853
- [Background] Barnsbee L, Barnett AG, Halton K, Nghiem S. Cost-effectiveness. In: Mechanical Circulatory and Respiratory Support. Elsevier; 2018:749-772. doi:10.1016/B978-0-12-810491-0.00024-2
- [Background] Sandelowski M. Sample size in qualitative research. Res Nurs Health. 1995 Apr;18(2):179-83. doi: 10.1002/nur.4770180211. PMID 7899572
- [Background] Boddy CR. Sample size for qualitative research. Qual Mark Res Int J. 2016;19(4):426-432. doi:10.1108/QMR-06-2016-0053
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006;3(2):77-101. doi:10.1191/1478088706qp063oa
- [Background] Familoni OB. An overview of stress in medical practice. Afr Health Sci. 2008 Mar;8(1):6-7. No abstract available. PMID 19357725
- [Background] Yeboah MA, Ansong MO, Antwi HA, Yiranbon E, Anyan F, Gyebil F. Determinants of Workplace Stress among Healthcare Professionals in Ghana: An Empirical Analysis. ResearchGate. 2014;Vol. 5(No. 4 [Special Issue]):140-151.
- [Background] Major B, Mendes WB, Dovidio JF. Intergroup relations and health disparities: a social psychological perspective. Health Psychol. 2013 May;32(5):514-24. doi: 10.1037/a0030358. PMID 23646834
- [Background] Chapman EN, Kaatz A, Carnes M. Physicians and implicit bias: how doctors may unwittingly perpetuate health care disparities. J Gen Intern Med. 2013 Nov;28(11):1504-10. doi: 10.1007/s11606-013-2441-1. Epub 2013 Apr 11. PMID 23576243
- [Background] Tincher MM, Lebois LA, Barsalou LW. Mindful attention reduces linguistic intergroup bias. Mindfulness (N Y). 2016 Apr;7(2):349-360. doi: 10.1007/s12671-015-0450-3. Epub 2015 Oct 15. PMID 27200110
- [Background] Gomez PP, Nelson AR, Asiedu A, Addo E, Agbodza D, Allen C, Appiagyei M, Bannerman C, Darko P, Duodu J, Effah F, Tappis H. Accelerating newborn survival in Ghana through a low-dose, high-frequency health worker training approach: a cluster randomized trial. BMC Pregnancy Childbirth. 2018 Mar 22;18(1):72. doi: 10.1186/s12884-018-1705-5. PMID 29566659
- [Background] Bluestone J, Johnson P, Fullerton J, Carr C, Alderman J, BonTempo J. Effective in-service training design and delivery: evidence from an integrative literature review. Hum Resour Health. 2013 Oct 1;11:51. doi: 10.1186/1478-4491-11-51. PMID 24083659
- [Background] Kujawski SA, Freedman LP, Ramsey K, Mbaruku G, Mbuyita S, Moyo W, Kruk ME. Community and health system intervention to reduce disrespect and abuse during childbirth in Tanga Region, Tanzania: A comparative before-and-after study. PLoS Med. 2017 Jul 11;14(7):e1002341. doi: 10.1371/journal.pmed.1002341. eCollection 2017 Jul. PMID 28700587
- [Background] Ndwiga C, Warren CE, Ritter J, Sripad P, Abuya T. Exploring provider perspectives on respectful maternity care in Kenya: "Work with what you have". Reprod Health. 2017 Aug 22;14(1):99. doi: 10.1186/s12978-017-0364-8. PMID 28830492
- [Background] Asefa A, Morgan A, Bohren MA, Kermode M. Lessons learned through respectful maternity care training and its implementation in Ethiopia: an interventional mixed methods study. Reprod Health. 2020 Jul 2;17(1):103. doi: 10.1186/s12978-020-00953-4. PMID 32615999
- [Background] Dzomeku VM, Boamah Mensah AB, Nakua EK, Agbadi P, Lori JR, Donkor P. Midwives' experiences of implementing respectful maternity care knowledge in daily maternity care practices after participating in a four-day RMC training. BMC Nurs. 2021 Mar 10;20(1):39. doi: 10.1186/s12912-021-00559-6. PMID 33691686
- [Background] Brown H, Hofmeyr GJ, Nikodem VC, Smith H, Garner P. Promoting childbirth companions in South Africa: a randomised pilot study. BMC Med. 2007 Apr 30;5:7. doi: 10.1186/1741-7015-5-7. PMID 17470267
- [Result] Khalil D. Violence against midwives in Cape Town. Afr J Midwifery Womens Health. 2009;3(1):37-40. doi:10.12968/ajmw.2009.3.1.39414
- [Result] WHO, UNICEF, UNFPA, The World Bank, United Nations Population Division. Trends in maternal mortality: 1990 to 2013. WHO. Published 2014. Accessed July 17, 2014. http://www.who.int/reproductivehealth/publications/monitoring/9789241503631/en/index.html
- [Derived] Afulani PA, Getahun M, Ongeri L, Aborigo R, Kinyua J, Ogolla BA, Okiring J, Moro A, Oluoch I, Dalaba M, Odiase O, Ouner JJ, Mendes WB, Walker D, Neilands TB. A cluster randomized controlled trial to assess the impact of the 'Caring for Providers to Improve Patient Experience' (CPIPE) intervention in Kenya and Ghana: study protocol. BMC Public Health. 2024 Sep 16;24(1):2509. doi: 10.1186/s12889-024-20023-9. PMID 39285405
- See also: Project website — https://personcenteredequitylab.ucsf.edu/projects#cpipe